CLINICAL TRIAL: NCT06608940
Title: A Phase Ib/II Study of BC3402, a Novel Anti-TIM3 Agent, in Combination With Tremelimumab Plus Durvalumab (STRIDE) in Advanced, Unresectable Hepatocellular Carcinoma
Brief Title: BC3402 w/ Tremelimumab + Durvalumab (STRIDE) in Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE5224
Record Dates: First submitted 2024-09-20; First posted 2024-09-23 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Hepato Cellular Carcinoma (HCC)
Keywords: liver cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BC3402 to tremelimumab plus durvalumab (Experimental): The study consists of two parts: a safety lead-in study part (Phase Ib) to confirm the tolerable dose (RP2D) of BC3402 in combination with T+D followed by an efficacy study part (Phase II) to evaluate preliminary efficacy of the study regimen in a single arm, two stage Minimax design. Note that participants who are treated at the RP2D in the Phase Ib study part will automatically be part of the Phase II study part.
  Interventions: Drug: BC3402; Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: BC3402 — BC3402, intravenous, 20 mg/kg, D1 and D15 of every 28 day cycle, continuous. BC3402 to be administered after completion of the infusion of durvalumab and/or tremelimumab on the days when BC3402 is to be administered with durvalumab and/or tremelimumab
Drug: Durvalumab — Durvalumab, intravenous, 1500 mg, every 4 weeks, continuous
Drug: Tremelimumab — Tremelimumab, intravenous, 300 mg, 1 dose on Cycle 1 Day 1

SUMMARY:
The purpose of this study is to test the safety and efficacy of an investigational (experimental) product called BC3402. This product is considered experimental because it is not approved by the U.S. Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
Brief Background/Rationale

Hepatocellular carcinoma (HCC) is the most common liver cancer and the fastest rising cause of cancer-related deaths in the U.S. Immune checkpoint inhibitors (ICIs) proved to be highly efficacious in HCC and the dual ICIs combination, tremelimumab plus durvalumab, is a standard front-line treatment for advanced and metastatic HCC. However, the response rate of the dual ICIs regimen is about 20% and participants invariably progress. There is a need for more efficacious treatment.

T cell immunoglobulin mucin-3 (TIM3) is highly expressed on multiple immune cells and plays a complex role in regulating immune responses and inducing immune tolerance. BC3402 is a TIM3 targeting inhibitory humanized IgG4 subtype monoclonal antibody which displays synergistic anti-tumor effects when combined with agents targeting PD1 and CTLA4 in preclinical tumor models as well as in the first in human (FIH) trial. Investigators hypothesize that the co-targeting of TIM3 will significantly increase the anti-tumor efficacy of dual targeting of PD1/PDL1 and CTLA4 axes in HCC and thus propose a clinical trial to investigate the efficacy of a novel triplet ICI combination of BC3402 plus the STRIDE regimen in participants with advanced, unresectable treatment-naïve HCC.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and any locally required authorization (eg, Health Insurance Portability and Accountability Act in the US, European Union [EU] Data Privacy Directive in the EU) obtained from the participant/legal representative prior to performing any protocol-related procedures, including screening evaluations.
* Confirmed HCC based on histopathological findings from tumor tissue.
* Must not have received prior systemic therapy for advanced, non-resectable HCC.
* Must not be eligible for locoregional therapy for unresectable HCC. For participants who progressed after locoregional therapy for HCC, locoregional therapy(including Transarterial chemoembolization (TACE) or Transarterial radioembolization (TARE)) must have been completed ≥28 days prior to the baseline scan for the current study.
* Barcelona Clinic Liver Cancer (BCLC) stage B (that is not eligible for locoregional therapy) or stage C.
* Child-Pugh Score class A.
* The Eastern Cooperative Oncology Group(ECOG) performance status of 0 or 1 at enrollment.
* Participants with Hepatitis B virus infection (as characterized by positive hepatitis B surface antigen [HBsAg], detectable HBV DNA, or hepatitis B core antibodies [anti-HBc Ab]) and are eligible for inclusion must be treated with antiviral therapy, per institutional practice, to ensure adequate viral suppression (HBV DNA ≤2000 IU/mL) prior to enrollment.

  o Note: HBV-positive participants must remain on antiviral therapy for the study duration and must continue therapy for 6 months after the last dose of study medication.
* Participants with Hepatitis C virus infection that are otherwise eligible for inclusion, must be confirmed by the presence of detectable HCV RNA or anti-HCV antibody upon enrollment (management of this disease is per local institutional practice).
* At least 1 measurable lesion, not previously irradiated and/or embolized, that can be accurately measured at baseline as ≥10 mm in the longest diameter (except lymph nodes, which must have a short axis ≥15 mm) with CT or MRI, and that is suitable for accurate repeated measurements as per RECIST 1.1 guidelines.
* Adequate organ and marrow function, as defined below. Criteria "a," "b," "c," and "f" cannot be met with transfusions, infusions, or growth factor support administered within 14 days of starting the first dose.

  1. Hemoglobin ≥9 g/dL
  2. Absolute neutrophil count ≥1000/μL
  3. Platelet count ≥75000/μL
  4. Total bilirubin (TBL) ≤2.0×ULN
  5. AST and ALT ≤5×ULN
  6. Albumin ≥2.8 g/dL
  7. International normalized ratio (INR) ≤1.6
  8. Calculated creatinine clearance ≥45 mL/minute as determined by Cockcroft-Gault (using actual body weight) or 24-hour urine creatinine clearance
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal participants.
* Must have body weight <100kg to be enrolled at the 20mg/kg dose level.

Exclusion Criteria:

* Any unresolved toxicity National Cancer Institute (NCI) Common Terminology Criteria for Adverse Event (CTCAE) Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria:
* Participants with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
* Participants with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Chair.
* Have received an investigational product or locoregional therapy within 28 days prior to the first dose of study drug(s).
* Any concurrent chemotherapy, study drug, or biologic or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (eg, hormone replacement therapy) is acceptable.
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
* Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 28 days of the first dose of study drug(s).
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of study drug(s). Note: Local surgery of isolated lesions for palliative intent is acceptable.
* History of allogeneic organ transplantation (eg, liver transplant).
* History of hepatic encephalopathy within past 12 months or requirement for medications to prevent or control encephalopathy (eg, no lactulose, rifaximin, etc if used for purposes of hepatic encephalopathy).
* Ascites that require ongoing paracentesis, within 6 weeks prior to the first scheduled dose of study drug(s), to control symptoms.
* Main portal vein thrombosis present on imaging.
* Active or prior documented GI variceal bleed or history of upper GI bleeding, ulcers, or esophageal varices with bleeding within 12 months; adequate endoscopic therapy according to institutional standards is required for participants with history of esophageal variceal bleeding or assessed as high risk for esophageal variceal by the treating investigator.
* Participant currently exhibits symptomatic or uncontrolled hypertension defined as diastolic blood pressure >90 mmHg or systolic blood pressure >140 mmHg.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). Participants without active disease in the last 5 years are excluded unless discussed with the Study Physician and considered appropriate for study participation. The following are exceptions to this criterion:
* Participants with vitiligo or alopecia
* Participants with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement
* Any chronic skin condition that does not require systemic therapy
* Participants with celiac disease controlled by diet alone
* Confirmed HBV infection must not be co-infected with HCV (as indicated by the absence of anti-HCV antibodies).
* Confirmed HCV infection must not be co-infected with HBV as defined by negative HBsAg. Participants with confirmed HCV infection who are negative for HBsAg, but positive for anti-HBc with detectable HBV DNA, are eligible but must be started on active antiviral therapy (for HBV) prior to enrollment to ensure adequate viral suppression (HBV DNA ≤2000 IU/mL).
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, Interstitial lung disease (ILD), serious chronic GI conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase the risk of incurring AEs, or compromise the ability of the participant to give written informed consent.
* History of another primary malignancy except for:
* Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of study drug(s) and of low potential risk for recurrence
* Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
* Adequately treated carcinoma in situ without evidence of disease
* History of leptomeningeal carcinomatosis.
* Brain metastases or spinal cord compression. Participants with suspected brain metastases at screening should have an MRI (preferred) or CT, each preferably with IV contrast of the brain prior to study entry.
* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
* History of active primary immunodeficiency.
* Active infection including tuberculosis (TB) (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), or human immunodeficiency virus (positive human HIV 1/2 antibodies).
* Current or prior use of immunosuppressive medication within 14 days before the first dose of study drug(s). The following are exceptions to this criterion:
* Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra-articular injection)
* Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
* Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication)
* Receipt of live attenuated vaccine within 30 days prior to the first dose of study drug(s). Note: Participants, if enrolled, should not receive live vaccine while receiving study drug(s) and up to 30 days after the last dose of study drug(s).
* Female participants who are pregnant or breastfeeding or male or female participants of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or 180 days after the last dose of durvalumab plus tremelimumab combination therapy. Not engaging in sexual activity, as per the participant's preferred and usual lifestyle, for the total duration of the treatment and washout periods is an acceptable practice.
* Prior randomization or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment.
* Participants who have received anti-PD-1, anti PD-L1, or anti CTLA-4 prior to the first dose of study drug(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate(ORR) per RECIST v1.1 | From registration up to 2 years post end of treatment(EOT) or study closure
  The ORR rate and 95% CI will be calculated.

SECONDARY OUTCOMES:
Duration of objective response | From registration up to 2 years post end of treatment(EOT) or study closure
  The duration of response will evaluated using waterfall plots where participants who continue to respond will be denoted by a circle.
Progression free survival(PFS), per RECIST v1.1 | From registration up to 2 years post end of treatment(EOT) or study closure
  PFS will be estimated via the Kaplan-Meier method.
Overall Survival(OS) | From registration up to 2 years post end of treatment(EOT) or study closure
  OS will be estimated via the Kaplan-Meier method.
Adverse events profile with AEs graded by the National Cancer Institute NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 | From registration up to 2 years post end of treatment(EOT) or study closure

CONTACTS AND LOCATIONS:
Locations (1):
- Case Comprehensive Cancer Center Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data included in the peer reviewed publication will be publicly available indefinitely. No raw data will be shared.
Access Criteria: A peer-reviewed publication will be made available according to the publishing journal's specifications. Cleveland Clinic Foundation personnel will not share study data apart from that which has been published publicly.
URL: https://pubmed.ncbi.nlm.nih.gov/